CLINICAL TRIAL: NCT03144089
Title: The Articulated Oral Airway as an Aid to Mask Ventilation, a Prospective Interventional, Non-Inferiority Study
Brief Title: The Articulated Oral Airway as an Aid to Mask Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ron Abrons (Other)
Responsible Party: Sponsor-Investigator, Ron Abrons, Assistant Professor of Anesthesiology, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201704829
Record Dates: First submitted 2017-04-17; First posted 2017-05-08 (Actual); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Mask Ventilation; Airway Obstruction Upper; Airway Management
Keywords: Morbid obesity; Obstructive sleep apnea; Mask ventilation; Upper airway obstruction
MeSH Terms: conditions — Obesity, Morbid; Sleep Apnea, Obstructive; Airway Obstruction

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, crossover design. All patients will receive both interventions during a single anesthetic, with the order of intervention being randomized.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Anesthesia facemasks will be opacified so that the clinical provider will be blinded to which oral airway (Guedel vs AOA) is being used and in what order. The patient will be anesthetized and thus blinded. The Investigator and Outcomes Assessor will only see video of the data on the anesthesia monitor (not the patient/device/etc) and will thus be blinded. The only individuals who will not be blinded are the Research Assistants who will not be involved in data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Guedel oral airway (Active Comparator): Each participant in the study will have both devices (GOA or AOA). The participants reported in this arm were randomized to receive the Guedel oral airway first and measurements were taken during breaths 6 through 10. After its removal the Articulated Oral Airway was inserted and measurements were repeated again during breaths 6 through 10.
  Interventions: Device: Guedel oral airway (active comparator)
- Articulated Oral Airway (Experimental): Each participant in the study will have both devices (GOA or AOA). The participants reported in this arm were randomized to receive the Articulated oral airway first and measurements were taken during breaths 6 through 10. After its removal the Guedel Oral Airway was inserted and measurements were repeated again during breaths 6 through 10.
  Interventions: Device: Articulated Oral Airway

INTERVENTIONS:
Device: Articulated Oral Airway — The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Other Names: AOA; Abrons AOA; Abrons Articulated Oral Airway
  Arms: Articulated Oral Airway
Device: Guedel oral airway (active comparator) — The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
  Arms: Guedel oral airway

SUMMARY:
The Articulating Oral Airway (AOA) is a novel oral airway which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The investigators hypothesize that, in patients with predictors for difficult mask ventilation, the AOA will be non-inferior to the Geudel oral airway in terms of expired tidal volumes.

DETAILED DESCRIPTION:
Difficult mask ventilation (MV) is common in the obese population and can result in patient morbidity and mortality. The Articulating Oral Airway (AOA) is a novel oral airway which actively displaces the tongue, allowing for a greater cross-sectional area for MV. The investigators hypothesize that, while using the same ventilatory pressure in neuromuscularly blocked patients with predictors for difficult mask ventilation, MV with an AOA will not result in smaller expired tidal volumes than MV with a similarly sized Guedel oral airway (GDA). In other words, the AOA will be non-inferior to the GDA in terms of expired tidal volumes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals demonstrating 2 or greater predictors of difficult mask ventilation (as listed below) who are scheduled for elective surgery with general anesthesia and asleep mask ventilation/orotracheal intubation utilizing long-acting neuromuscular blockade.
* Predictors of difficult mask ventilation i) Age > 55 years ii) BMI > 30kg/m2 iii) Beard iv) Lack of teeth v) History of snoring

Exclusion Criteria:

* Documented history of impossible mask ventilation
* Planned omission of mask ventilation ('rapid-sequence induction,' etc.)
* Planned omission of long-acting paralytics
* Need for awake airway management
* Need for emergent airway protection
* Presence of oropharyngeal anatomic abnormalities
* Distance from the maxillary incisors to the angle of the mandible <11cm
* <18 years of age
* Known pregnant state
* Current incarceration
* Refusal to be involved in the study

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-07-11 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2019-02-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron O Abrons, MD, Principal Investigator — The University of Iowa Hospitals and Clinics
Locations (1):
- The University of Iowa Hospital, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koga K, Sata T, Kaku M, Takamoto K, Shigematsu A. Comparison of no airway device, the Guedel-type airway and the Cuffed Oropharyngeal Airway with mask ventilation during manual in-line stabilization. J Clin Anesth. 2001 Feb;13(1):6-10. doi: 10.1016/s0952-8180(00)00228-2. PMID 11259887
- [Background] Langeron O, Masso E, Huraux C, Guggiari M, Bianchi A, Coriat P, Riou B. Prediction of difficult mask ventilation. Anesthesiology. 2000 May;92(5):1229-36. doi: 10.1097/00000542-200005000-00009. PMID 10781266
- [Background] Kheterpal S, Han R, Tremper KK, Shanks A, Tait AR, O'Reilly M, Ludwig TA. Incidence and predictors of difficult and impossible mask ventilation. Anesthesiology. 2006 Nov;105(5):885-91. doi: 10.1097/00000542-200611000-00007. PMID 17065880
- [Background] Kheterpal S, Martin L, Shanks AM, Tremper KK. Prediction and outcomes of impossible mask ventilation: a review of 50,000 anesthetics. Anesthesiology. 2009 Apr;110(4):891-7. doi: 10.1097/ALN.0b013e31819b5b87. PMID 19293691
- [Derived] Abrons RO, Ten Eyck P, Sheffield ID. The Articulated Oral Airway as an aid to mask ventilation: a prospective, randomized, interventional, non-inferiority study. BMC Anesthesiol. 2021 Mar 29;21(1):94. doi: 10.1186/s12871-021-01315-8. PMID 33781212

RESULTS

PARTICIPANT FLOW:
Groups:
- Guedel Oral Airway Placed First: This group is randomized to receive the Guedel oral airway first and the Articulated Oral Airway second
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
- Articulated Oral Airway Placed First: This group is randomized to receive the Articulated Oral Airway first and the Guedel oral airway second
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
Period: Overall Study
Arm/Group | Guedel Oral Airway Placed First | Articulated Oral Airway Placed First
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Guedel Oral Airway Placed First | Articulated Oral Airway Placed First | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 15 | 34
  >=65 years | 9 | 13 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 16 | 19 | 35
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56
BMI [Median (Full Range); unit: kg/m^2] | 34.8 [31.0 to 39.0] | 36.1 [33.0 to 40.0] | 35.4 [31.0 to 40.0]

OUTCOME MEASURES:

1. Primary Outcome: Expiratory Tidal Volume (Breaths 6-10)
Description: Measured expiratory tidal volume (from video of anesthesia monitor). Each participant had measurements collected during breaths number 6-10 after the insertion of each oral airway (GOA or AOA) with the order of first treatment randomized. The average expiratory tidal volumes reported were weight standardized per kilogram of participant's body weight, meaning the expiratory measurements were divided by the participant's weight (kg). A total of 56 patients were enrolled and randomized--28 received the Guedel Oral Airway first and 28 received the Articulated Oral Airway first. The average expiratory values are reported as outlined in table below:
  Guedel inserted first AOA inserted first Guedel inserted second AOA inserted second
Time Frame: Measured immediately after placement of each oral airway; an average of 2-5 minutes.
Measure: Mean (95% Confidence Interval); unit: ml/kg
Groups:
- Guedel Oral Airway: This group is randomized to receive the Guedel oral airway first and the Articulated Oral Airway second
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
- Articulated Oral Airway: This group is randomized to receive the Articulated Oral Airway first and the Guedel oral airway second
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
Arm/Group | Guedel Oral Airway | Articulated Oral Airway
Number analyzed (Participants) | 28 | 28
ml/kg
  First intervention-breaths 6 through 10 | 4.46 [3.86 to 5.07] | 3.21 [2.62 to 3.79]
  Second intervention-breaths 6 through 10 | 3.12 [2.54 to 3.70] | 3.48 [2.87 to 4.08]

2. Secondary Outcome: Inspiratory Tidal Volume (Breaths 6-10)
Description: Measured inspiratory tidal volume (from video of anesthesia monitor). Each participant had measurements collected during breaths number 6-10 after the insertion of each oral airway (GOA or AOA) with the order of first treatment randomized. The average inspiratory tidal volumes reported were weight-standardized per kilogram of participant's body weight, meaning the inspiratory measurements were divided by the participant's weight (kg). A total of 56 patients were enrolled and randomized--28 received the Guedel Oral Airway first and 28 received the Articulated Oral Airway first. The average inspiratory values are reported as outlined in table below:
  Guedel inserted first AOA inserted first Guedel inserted second AOA inserted second
Time Frame: Measured immediately after placement of each oral airway; an average of 2-5 minutes.
Measure: Mean (95% Confidence Interval); unit: ml/kg
Arm/Group | Guedel Oral Airway | Articulated Oral Airway
Number analyzed (Participants) | 28 | 28
ml/kg
  First intervention-breaths 6 though 10 | 6.37 [5.35 to 7.40] | 5.7 [4.71 to 6.68]
  Second intervention-breaths 6 through 10 | 5.83 [4.84 to 6.82] | 6.72 [5.70 to 7.75]

3. Secondary Outcome: Immediate Oropharyngeal Trauma From Oral Airway Randomized to be Placed First
Description: After the first oral airway device was removed, it was visually inspected for the presence of blood and is reported as the number of subjects where blood was visualized on the initial airway device..
Time Frame: Measured immediately after removal of first oral airway and before placing the second oral airway
Measure: Number; unit: Devices with blood
Arm/Group | Guedel Oral Airway Placed First | Articulated Oral Airway Placed First
Number analyzed (Participants) | 28 | 28
Devices with blood | 3 | 0

ADVERSE EVENTS:
Time Frame: Day of surgical procedure.
Groups:
- Guedel Oral Airway: This group is randomized to receive the Guedel oral airway first and data recorded. The airway was removed and followed by insertion of the Articulated Oral Airway second and data recorded.
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
- Articulated Oral Airway: This group is randomized to receive the Articulated Oral Airway first and data recorded. The airway was removed and followed by insertion the Guedel oral airway second and data recorded.
  Articulated Oral Airway: The AOA is a novel device which actively displaces the tongue, allowing for a greater cross-sectional area for mask ventilation. The AOA will be evaluated for efficacy of mask ventilation.
  Guedel oral airway (active comparator): The Guedel oral airway is a standard oral airway commonly used to facilitate mask ventilation. The Guedel oral airway will be evaluated for efficacy of mask ventilation.
Arm/Group | Guedel Oral Airway | Articulated Oral Airway
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03144089/Prot_SAP_003.pdf
  • Informed Consent Form (2021-05-16): https://cdn.clinicaltrials.gov/large-docs/89/NCT03144089/ICF_004.pdf